CLINICAL TRIAL: NCT05916625
Title: Exploratory Study of the Expression of the Serotonergic 5-HT4 Receptor in Parkinson's
Brief Title: Exploratory Study of the Expression of the Serotonergic 5-HT4 Receptor in Parkinson's Disease
Acronym: PARK 5-HT4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL22_0953
Record Dates: First submitted 2023-04-12; First posted 2023-06-23 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
Keywords: serotonergic 5-HT4 receptor; radiotracer
MeSH Terms: conditions — Parkinson Disease | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pet scan with the specific radioligand [11C]SB207145 (Experimental): The following examen are added by the study :
  neuropsychologic consultation PET scan MRI biological sample Questionnaires
  Interventions: Other: neuropsychological assessment; Other: biological sample; Procedure: medical imagery

INTERVENTIONS:
Other: neuropsychological assessment — a consultation to assess cognitive and psycho-behavioral functions with questionnaires
Other: biological sample — 10 mL intravenous whole blood collection in EDTA tube
Procedure: medical imagery — Pet scan with the specific radioligand [11C]SB207145 and MRI

SUMMARY:
The research aim to study in detail the motor, cognitive and affective modifications of Parkinsonian patients (compared to control subjects) at a moderate stage of the disease and to analyze by positron emission tomography (PET) imaging with the specific radioligand [11C]SB207145 the expression levels of this 5-HT4 receptor. At the same time, the study will monitor the impact of the 5-HTTLPR polymorphisms of Serotonin Transporter (SERT) and Brain-derived neurotrophic factor (BDNF) Val66Met on the expression of the 5-HT4 receptor in subjects.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman : Age between ≥ 50 and ≤ 85 years old
* For women: postmenopausal
* Affiliated to a social security scheme or similar;
* Having given written consent to participate in the free and informed study.
* Level of study: ≥ 6 years of schooling
* only for healthy volunteer : No history of neurological or psychiatric disease
* Only for patient : Having a clinically established or probable diagnosis of Parkinson's disease according to the criteria defined by the Movement Disorder Society at a Hoehn and Yahr stage ≤ 3 (in on dopa conditions) and a duration of evolution of the disease between 2 and 8 years.
* Only for patient : Having a MoCA (Montreal Cognitive Assessment) ≥ 20/30.

Exclusion Criteria:

* Diagnosis other than Parkinson's disease ( for patient only)
* Treated with specific serotonin inhibitors (SSRIs), specific noradrenaline inhibitors (SNRIs), tricyclic antidepressants, monoamine oxidase inhibitors (MAOIs) and neuroleptics in the last 3 months
* Use of recreational drugs interfering with the serotonergic system (ecstasy, MDMA) or opioids (cannabis, opiates) in the last 3 months or chronic use
* Contraindication to magnetic resonance imaging (MRI) or positron emission tomography (PET)
* Participation in the last year to a study using ionizing radiation or concomitant participation in another research project involving the human being that may interfere with the results or the conclusions of this study
* Exceeding the annual amount of compensation authorized for participation in research protocols
* Deprivation of liberty by judicial or administrative decision, person subject to a legal protection measure
* BMI ≥ 35kg/m2
* Presence of depression (BDI-2 score ≥21), anxiety (Parkinson Anxiety Scale (PAS) score ≥14) or apathy (STARKSTEIN score ≥14) - (for healthy volunteers only)
* Cognitive impairment (MOCA score ≤26) (for healthy volunteers only)
* Current or past neurological or psychiatric pathology (for healthy volunteers only)
* Serious and progressive medical pathology
* Current or past dependence on any addictive substance according to DSM-V (The Diagnostic and Statistical Manual of Mental Disorders) criteria (alcohol, cannabis, hallucinogens, inhalants, opiates, sedatives, stimulants), except tobacco and caffeine. (for healthy volunteers only)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Comparison of the expression of the 5-HT4 receptor between patients with mild to moderate Parkinson's disease to age-matched healthy controls | During MRI procedure
  difference in the tracer [11C]SB207145 's binding, the specific binding of the tracer will be calculated for each voxel with respect to a reference zone (the white matter of the cerebellum).

SECONDARY OUTCOMES:
Description of 5-HT4 alterations related to motor symptoms | During MRI procedure
  Relationship between the level of expression of the tracer and the clinical scores on the motor questionnaires
Description of 5-HT4 alterations related to non-motor symptoms | During MRI procedure
  Relationship between the level of expression of the tracer and the clinical scores on the non-motor questionnaires
Description of 5-HT4 alterations related to cognitive symptoms | During MRI procedure
  Relationship between the level of expression of the tracer and the clinical scores on the cognitive questionnaires
Description of 5-HT4 alterations related to psychobehavioral symptoms | During MRI procedure
  Relationship between the level of expression of the tracer and the clinical scores on the psychobehavioral questionnaires
Description of 5-HT4 alterations related to SERT polymorphism data | During MRI procedure
  Relationship between the level of expression of the tracer and SERT polymorphism data (5-HTTLPR polymorphism, evaluated as presence/absence)
Description of 5-HT4 alterations related to BDNF polymorphism data | During MRI procedure
  Relationship between the level of expression of the tracer and BDNF polymorphism data (Val66Met rs6265 polymorphism, evaluated as presence/absence)

CONTACTS AND LOCATIONS:
Overall Officials: Jing XIE, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - CERMEP, Bron
  - Hôpital des Charpennes Centre de Recherche Clinique "Vieillissement-Cerveau-Fragilité", Lyon